CLINICAL TRIAL: NCT03736824
Title: Correlation of Endoscopic Findings and Symptoms in Patients Undergoing the First Upper Gastrointestinal Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, Shanghai Jiao Tong University School of Medicine
Other Study IDs: rjyy20181021
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Symptoms and Signs; Malignancy; Ulcer Peptic
MeSH Terms: conditions — Signs and Symptoms; Neoplasms; Peptic Ulcer | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endoscopy — All endoscopy was performed by qualified gastroenterologists or endoscopic physicians in Renji hospital,Shanghai Jiaotong University School of Medicine.

SUMMARY:
Endoscopy is the best means of finding early stage of upper gastrointestinal diseases, especially early cancer and benign ulcers. Currently, most people still undergo upper gastrointestinal endoscopy due to discomfort, rather than a regular physical examination at a certain age. This study prospectively investigated the reason for undergoing the first upper gastrointestinal endoscopy in patients and found the correlation of endoscopic findings and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing the first upper gastrointestinal endoscopy.

Exclusion Criteria:

* The patients had previously performed endoscopy and any esophageal, gastric or duodenal surgery.
* The patients couldn't complete the questionnaire survey under the guidance of physicians at the appointment of the upper gastrointestinal endoscopy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing the first upper gastrointestinal endoscopy were collected from January 2018 to December 2018 in Renji Hospital, Shanghai Jiaotong University School of Medicine.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of endoscopic findings and symptoms | Within two weeks after receiving the survey
  survey

SECONDARY OUTCOMES:
The proportion of various symptoms in patients undergoing the first upper gastrointestinal endoscopy | Within two weeks after receiving the survey
The proportion of different upper gastrointestinal diseases | Within two weeks after receiving the survey
  Diagnosis of upper gastrointestinal disease combined with endoscopic findings and pathological diagnosis.
The infection rate of Helicobacter Pylori | Within two weeks after receiving the survey
  H. pylori infection was determined by any two of positive outcome of the breath test, rapid urease test and histology.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, Study Director — School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided